CLINICAL TRIAL: NCT05113979
Title: Early Feasibility Study to Evaluate the Safety and Effectiveness of the AccuraSee for Secondary Implantation in the Capsular Bag to Correct Residual Refractive Errors of Previous Cataract Surgery
Brief Title: Early Feasibility Study to Evaluate the AccuraSee in Correcting Residual Refractive Errors After Cataract Surgery
Status: Completed | Type: Interventional
Sponsor: OnPoint Vision Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIIPCL-018
Record Dates: First submitted 2021-08-04; First posted 2021-11-09 (Actual); Results first posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Refractive Errors
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Intervention Model Description: Treatment with AccuraSee Intraocular Pseudophakic Contact Lens (IOPCL) at least 6-months after cataract surgery with Bausch and Lomb Model LI61A0 and LI61SE
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (1):
- IOPCL (Experimental): Intraocular Pseudophakic Contact Lens (IOPCL) with +3.0D add
  Interventions: Device: AccuraSee IOPCL with +3.0D add

INTERVENTIONS:
Device: AccuraSee IOPCL with +3.0D add — The IOPCL (intraocular pseudophakic contact lens) consists of a 4.5mm diameter optic. All subjects will receive a +3.0 power regardless of diopter power based on IOL Master. This IOPCL will be coupled to a Bausch and Lomb Model LI61SE or LI61AO intraocular lens to correct residual refractive errors after cataract surgery.

SUMMARY:
To determine if the intraocular pseudophakic contact lens (IOPCL), referred to as the AccuraSee, corrects residual refractive errors after cataract surgery using a plus powered lens in subjects with ocular pathology previously implanted with a Bausch and Lomb LI61AO or LI61SE monofocal posterior chamber intraocular lens (PCIOL) and to confirm its positional stability and adherence relative to the PCIOL.

DETAILED DESCRIPTION:
This will be a 12-month study in which a maximum of 10 pseudophakic patients from three clinical sites will be enrolled. All enrolled subjects will receive an AccuraSee IOPCL with +3.0D add to correct residual refractive errors identified after cataract surgery.

The primary objective of this study is to determine the stability of the AccuraSee IOPCL to successfully adhere to a pseudophakic intraocular lens (PCIOL) without rotation or slippage.

The secondary objective of this study is to determine if the AccuraSee IOPCL can successfully correct refractive errors in subjects previously implanted with a Bausch and Lomb LI61AO and LI61SE monofocal intraocular lens.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have already had cataract surgery with a Bausch and Lomb monofocal intraocular lens model LI61AO (with lens power from 18.0 diopters (D) to 23.0 D) or model LI61SE monofocal intraocular lens (with a lens power between from18.0 D and 23.0 D), clearly evidenced by photographic documentation with one of the following: (1) patient medical record, (2) clinic chart with labeling attached, (3) surgical record with labeling attached, or (4) patient identification card with make, model, power, and serial number.
* Able to comprehend and sign a statement of informed consent.
* Willing and able to complete all required postoperative visits.
* Subjects who's baseline manifest refraction spherical equivalent (MRSE) is between -0.5D and +3.0D
* Best corrected visual acuity 20/80 or worse.
* Subjects with ≤1.0D 5D of refractive corneal cylinder
* Subjects willing to abstain from pursuing any other surgical vision-correcting procedures for the duration of the study.
* Subject must be at least 22 years or older.

Exclusion Criteria:

* Subjects who have already had cataract surgery with a Toric or multifocal Intraocular Lens.
* Subjects who have already had cataract surgery with a Bausch and Lomb monofocal intraocular lens model LI61AO (with a lens power below 18.0 D and greater than 23.0 D) or model LI61SE (with a lens power below 18.0 D and greater than 22.5 D).
* Subjects who were treated with an IOL off-label.
* Subjects who have MRSE of less than 1.0 Diopter (+1.0 to -1.0 D) and more than +3.0D
* Subjects who have more than 1.5D of refractive corneal cylinder
* Subjects whose continuous curvilinear capsulorhexis was less than 5mm or more than 6.0 mm in size at the time of IOL surgery.
* Subjects who had cataract surgery less than 6 months from the planned date of the IOPCL surgery.
* Subjects with anterior capsule fibrosis and phimosis that in the opinion of the investigator may confound the outcome or increase the risk to the subject.
* Acute, chronic or uncontrolled systemic or ocular disease that in the opinion of the investigator would increase the operative risk or confound the outcome(s) of the study.
* Any corneal abnormality, other than regular corneal astigmatism that in the opinion of the investigator would confound the outcome(s) of the study.
* Clinically severe corneal dystrophy (e.g., epithelial, stromal, or endothelial dystrophy).
* Microphthalmos.
* Previous retinal detachment.
* Recurrent severe anterior or posterior segment inflammation of unknown etiology.
* Iris neovascularization.
* Uncontrolled glaucoma.
* Aniridia.
* Optic nerve atrophy.
* Damaged or incomplete zonules.
* Known history of pseudoexfoliation.
* Medications that, in the opinion of the investigator, may confound the outcome or increase the risk to the subject (tamsulosin hydrochloride (Flomax)) or other medications with similar side effects (floppy iris syndrome).

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2022-09-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Vision Institute, Bloomington, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited and enrolled (consented) at three private medical clinics between March 9, 2020 and November 2, 2021.
Pre-assignment Details: Of the 12 consented participants, 10 met all study eligibility criteria and were enrolled into the study. Nine met intraoperative eligibility and were treated with the AccuraSee intraocular pseudophakic contact lens (IOPCL) with +3.0D add.
Groups:
- Intent-to-Treat: All eligible, enrolled subjects in which the AccuraSee intraocular pseudophakic contact lens (IOPCL) with +3.0D add implantation was attempted
Period: Overall Study
Arm/Group | Intent-to-Treat
Started | 10
Completed | 7
Not Completed | 3
Not completed — Death | 2
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Intent to Treat (ITT) - All patients that were enrolled and attempted implantation of the Intraocular Pseudophakic Contact Lens (IOPCL)
Groups:
- Intent-to-Treat: All eligible, enrolled subjects in which the AccuraSee intraocular pseudophakic contact lens (IOPCL)with +3.0D add implantation was attempted
Arm/Group | Intent-to-Treat
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: Years] — Equal to or greater than 22 years of age.
  Years | 79.3 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Subjects With Stable Manifest Refraction Spherical Equivalent (MRSE)
Description: Proportion of subjects (≥ 50%) able to achieve MRSE stability within ±0.5D within two consecutive postoperative visits at 1 month or later visits.
Time Frame: Assessed all postoperative consecutive visit pairings beginning with 1 month visit (1 month to 4 months; 4 months to 1 year); reported for "Postoperative period between 1 month and 1 year"
Population: All treated subjects with two or more consecutive postoperative visits
Measure: Number; unit: Subjects
Groups:
- Subjects Treated With AccuraSee IOPCL With +3.0D Add: All subjects treated with AccuraSee intraocular pseudophakic contact lens (IOPCL) with +3.0D add
Arm/Group | Subjects Treated With AccuraSee IOPCL With +3.0D Add
Number analyzed (Participants) | 8
Subjects | 7

2. Primary Outcome: Subjects With Successful Delivery of AccuraSee IOPCL
Description: Successful delivery of the AccuraSee IOPCL is defined as: 1) No capsular tear; 2) Visualized centration between the PCIOL and the IOPCL; 3) No visible damage to either the PCIOL or the IOPCL; and 4) Uniform leaflet coverage of all IOPCL haptic tabs
Time Frame: 7-14 days visit
Population: All treated subjects that completed the 7-14 days visit
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects Treated With AccuraSee IOPCL With +3.0D Add
Number analyzed (Participants) | 9
Participants
  Capsular tear: No | 9
  Capsular tear: Yes | 0
  Visualized centration between the PCIOL and IOPCL: No | 0
  Visualized centration between the PCIOL and IOPCL: Yes | 9
  Visible damage to either the PCIOL or the IOPCL: No | 9
  Visible damage to either the PCIOL or the IOPCL: Yes | 0
  Uniform leaflet coverage of all IOPCL haptic tabs: No | 0
  Uniform leaflet coverage of all IOPCL haptic tabs: Yes | 9

3. Primary Outcome: Long Term Adherence and Positional Stability: Number of Participants With Greater or Less Than +/- 10 Microns Change in Gap Between the Pseudophakic Intraocular Lens and AccuraSee Intraocular Pseudophakic Contact Lens
Description: Safety Endpoint: Minimal change in uniformity of the gap between the pseudophakic intraocular lens (PCIOL) and AccuraSee intraocular pseudophakic contact lens (IOPCL), between 30-60 days and 120-180 days, as determined by ultrasound biomicroscopy (UBM) measurements. Minimal change is defined as +/- 10 microns.
Time Frame: Assessed at 30-60 days visit and 120-180 days visit, 120-180 days visit reported
Population: All treated subjects that completed the 30-60 days visit and 120-180 days visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects Treated With AccuraSee IOPCL With +3.0D Add
Number analyzed (Participants) | 8
Participants
  Gap with less than +/- 10 microns change | 8
  Gap with greater than +/- 10 microns change | 0

4. Other Pre Specified Outcome: Change in UCDVA From Baseline
Description: Change in Uncorrected Distance Visual Acuity (UCDVA) from Baseline measured in lines (5 letters) on ETDRS (Early Treatment Diabetic Retinopathy Study)
Time Frame: Baseline and 330-420 days
Population: All subjects that completed the 330-420 days visit
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects Treated With AccuraSee IOPCL With +3.0D Add
Number analyzed (Participants) | 7
Participants
  > 2 lines gained | 0
  2 lines gained | 2
  1 line gained | 0
  No change | 4
  1 line loss | 0
  2 lines lost | 0
  > 2 lines lost | 1

ADVERSE EVENTS:
Time Frame: 12-Months
Description: Any untoward or unfavorable medical occurrence, unintended disease or injury, whether or not related to the investigational medical device. All intent-to-treat (ITT) subjects, which underwent IOPCL implantation attempt, were evaluated for adverse events.
Arm/Group | Intent-to-Treat
All-Cause Mortality (participants affected / at risk) | 2/10
Serious Adverse Events (participants affected / at risk) | 2/10
Other Adverse Events (participants affected / at risk) | 2/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intent-to-Treat (N=10)
Death secondary to kidney failure (Renal and urinary disorders) | 1 (1)
Death (Cardiac disorders) | 1 (1) — Death due to natural causes
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intent-to-Treat (N=10)
Unseated haptic tab (Eye disorders) | 1 (1) — One or more AccuraSee IOPCL haptic tabs not securely attached to the PCIOL
Failure to implant IOPCL (Eye disorders) | 1 (1) — Failure to implant IOPCL due to intraoperative discovery of phacodonesis (pre-existing)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol: Clinical Protocol (2021-04-08): https://cdn.clinicaltrials.gov/large-docs/79/NCT05113979/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-08): https://cdn.clinicaltrials.gov/large-docs/79/NCT05113979/SAP_003.pdf
  • Informed Consent Form: Informed consent document (2021-07-16): https://cdn.clinicaltrials.gov/large-docs/79/NCT05113979/ICF_002.pdf